CLINICAL TRIAL: NCT04461834
Title: Accuracy of the RIVA Digital Blood Pressure Measurement App After Initial Calibration and After 24 Hours in a General Population - a Pilot Study
Brief Title: Accuracy of the RIVA Digital Blood Pressure Measurement App - a Pilot Study
Status: Completed | Type: Observational
Sponsor: CSEM Centre Suisse d'Electronique et de Microtechnique SA - Recherche et Developpement (Industry)
Collaborators: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: RIVA_Basel
Record Dates: First submitted 2020-07-02; First posted 2020-07-08 (Actual); Last update posted 2020-10-01 (Actual); Status verified 2020-09

CONDITIONS: Blood Pressure
Keywords: Blood Pressure; RIVA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this pilot study is to test the accuracy of the RIVA Digital Blood Pressure Measurement App with and without initial calibration. Additionally, accuracy of the Blood Pressure Measurement 24 hours after calibration will also be tested.

DETAILED DESCRIPTION:
Conventional blood pressure measurements (BPM) using a cuff-based device are actually gold standard of BPM in clinical practice. Due to availability and patient comfort, the number of such BPM is limited. Considering the large number of people using smartphones, app-based measurements and screening procedures have the potential to increase the availability of BPM and improve blood pressure control, but a prerequisite of the use of these alternative BPM methods is accuracy.

The aim of this pilot study is to test the accuracy of the RIVA Digital Blood Pressure Measurement App with and without initial calibration. Additionally, accuracy of the BPM 24 hours after calibration will also be tested.

Before mounting the 24h-Blood Pressure (BP) monitor, a set of 11 BPM will be taken, starting with a conventional BPM using a Welch Allyn Connex® Spot Monitor, then alternating to the app, leading to 6 possible pairs of comparison. The next day, without another calibration of the app, we will take another 3 pairs of comparison (7 alternating measurements, starting with a conventional measurement). Examinators are blinded for the results of the app measurements. The app automatically sends the data of the BPM to RIVA Digital, where the results measured by the app will be processed. The staff of RIVA Digital are blinded to the conventional BPM results.

Number of Participants: 50 consecutive patients will be included in the study.

Statistical analyses: Both BPM procedures are analyzed for correlation and accuracy.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing a 24h-ambulatory blood pressure measurement

Exclusion Criteria:

* age < 18 years
* impossibility to sign informed consent
* physical restrictions to Blood Pressure Measurement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AIl patients undergoing a 24h-ambulatory blood pressure measurement are eligible.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-06-25 (Actual); Primary Completion 2020-09-24 (Actual); Study Completion 2020-09-24 (Actual)

PRIMARY OUTCOMES:
Data statistical analysis | 1 year
  Both Blood Pressure Measurement procedures are analysed for correlation and accuracy

CONTACTS AND LOCATIONS:
Overall Officials: Michael Mayr, PD Dr., Principal Investigator — University Hospital of Basel
Locations (1):
- University Hospital of Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No